CLINICAL TRIAL: NCT01239589
Title: European Study to Describe Hospital Stay in Patients Admitted for Acute Bipolar Manic Episodes Treated With Immediate Release Quetiapine or Extended Release Quetiapine
Brief Title: European Study to Describe Hospital Stay in Patients Admitted for Acute Bipolar Manic Episodes
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Medical Science Director, AstraZeneca
Other Study IDs: NIS-NEU-SER-2010/1
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Acute Bipolar Manic Episode
Keywords: Patients admitted as for an acute bipolar manic episode; Description of management patterns and hospital stay in patients admitted for acute bipolar manic episode and treated with either quetiapine IR or quetiapine XR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: patients admitted as for an acute bipolar manic episode and treated with quetiapine IR
- 2: patients admitted as for an acute bipolar manic episode and treated with quetiapine XR

SUMMARY:
This study is being carried out to find out how patients suffering from the acute manic phase of bipolar disease are currently managed with Quetiapine Immediate Release (IR) or Quetiapine Extended Release (XR) in the hospital setting in real life practice, including length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Bipolar Disorder (ICD-10).
* Admitted for acute bipolar manic episode from 1st October 2009 to 1st October 2010
* Patients treated with quetiapine IR or quetiapine XR during the hospitalization period.

Exclusion Criteria:

* Patients in which BD is not the main reason for hospitalization
* Patients admitted for acute bipolar mania episodes but finally diagnosed with mixed or bipolar disorder not otherwise specified (NOS) episodes
* Patients receiving both quetiapine IR and XR during the same hospitalization period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Bipolar Disorder (ICD-10).admitted due to a acute manic episode and treated with quetiapine IR or quetiapine XR during the hospitalization period
Sampling Method: Probability Sample
Enrollment: 1280 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay

SECONDARY OUTCOMES:
Use of resources
Treatments used
Demographics

CONTACTS AND LOCATIONS:
Locations (86):
- Belgium (13):
  - Research Site, Assebroek, Belgium
  - Research Site, Bertrix, Belgium
  - Research Site, Bruges, Belgium
  - Research Site, Ghent, Belgium
  - Research Site, Godinne, Belgium
  - Research Site, Ixelles-Elsene, Belgium
  - Research Site, Koksijde, Belgium
  - Research Site, Malle, Belgium
  - Research Site, Marchienne-au-Pont, Belgium
  - Research Site, Montignies-sur-Sambre, Belgium
  - Research Site, Ottignies, Belgium
  - Research Site, Overpelt, Belgium
  - Research Site, Roeselaere, Belgium
- Croatia (2):
  - Research Site, Zagreb, City of Zagreb
  - Research Site, Split, Split
- Denmark (4):
  - Research Site, Augustenborg, Augustenborg
  - Research Site, Bispebjerg, Bispebjerg
  - Research Site, Br�nderslev, Br�nderslev
  - Research Site, Odense, Odense
- Finland (4):
  - Research Site, Helsingin Kaupunki, Helsingin Kaupunki
  - Research Site, Jyv�skyl�, Jyv�skyl�
  - Research Site, Kellokoski, Kellokoski
  - Research Site, Ekenäs, Tammisaari
- Germany (12):
  - Research Site, Ulm, Baden-W�rttemberg
  - Research Site, Cham, Bavaria
  - Research Site, Neu�tting, Bavaria
  - Research Site, Regensburg, Bavaria
  - Research Site, Wasserburg am Inn, Bavaria
  - Research Site, W�rzburg, Bavaria
  - Research Site, Bielefeld, Lower Saxony
  - Research Site, Hildesheim, Lower Saxony
  - Research Site, Liebenburg, Lower Saxony
  - Research Site, Greifswald, Mecklenburg-Vorpommern
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Berlin, State of Berlin
- Italy (17):
  - Research Site, Ascoli Piceno, Ascoli Piceno
  - Research Site, Bologna, Bologna
  - Research Site, Ceglie Messapica, Brindisi
  - Research Site, San Pietro Vernotico, Brindisi
  - Research Site, Lamezia Terme, Catanzaro
  - Research Site, Cosenza, Cosenza
  - Research Site, Cuneo, Cuneo
  - Research Site, Ferrara, Ferrara
  - Research Site, Foggia, Foggia
  - Research Site, Loc. S. Marciano (Sora), Frosinone
  - Research Site, S. Agata Militello, Messina
  - Research Site, Mestre, Mestre
  - Research Site, Pisa, Pisa
  - Research Site, Roma, Roma
  - Research Site, Sassari, Sassari
  - Research Site, Teramo, Teramo
  - Research Site, Conegliano, Treviso
- Turkey (Türkiye) (16):
  - Research Site, Adana, Adana
  - Research Site, Ankara, Ankara
  - Research Site, Ayd?n, Ayd?n
  - Research Site, Bolu, Bolu
  - Research Site, Diyarbakır, Diyarbakır
  - Research Site, Elâzığ, Elâzığ
  - Research Site, Erzurum, Erzurum
  - Research Site, Istanbul, Istanbul
  - Research Site, Kayseri, Kayseri
  - Research Site, Konya, Konya
  - Research Site, Manisa, Manisa
  - Research Site, Samsun, Samsun
  - Research Site, Sivas, Sivas
  - Research Site, Trabzon, Trabzon
  - Research Site, Zonguldak, Zonguldak Province
  - Research Site, Sanliurfa, Şanlıurfa
- United Kingdom (18):
  - Research Site, Bury St Edmunds, Bury Saint Edmunds
  - Research Site, Winsford, Cheshire
  - Research Site, Coventry, Coventry
  - Research Site, Hull, Hull
  - Research Site, Dartford, Kent
  - Research Site, Leeds, Leeds
  - Research Site, Leicester, Leicester
  - Research Site, Ealing, London
  - Research Site, London, London
  - Research Site, Prescot, Merseyside
  - Research Site, Newcastle upon Tyne, Newcastle (Upon Tyne)
  - Research Site, Norwich, Norfolk
  - Research Site, Taunton, Somerset
  - Research Site, Cannock, Staffordshire
  - Research Site, Chertsey, Surrey
  - Research Site, Wolverhampton, West Midlands
  - Research Site, Pulborough, West Sussex
  - Research Site, Bradford, Yorkshire

REFERENCES:
- [Derived] Karamustafalioglu O, Reif A, Atmaca M, Gonzalez D, Moreno-Manzanaro M, Gonzalez MA, Medina E, Bellomo A. Hospital stay in patients admitted for acute bipolar manic episodes prescribed quetiapine immediate or extended release: a retrospective non-interventional cohort study (HOME). BMC Psychiatry. 2014 Aug 31;14:246. doi: 10.1186/s12888-014-0246-3. PMID 25174996